CLINICAL TRIAL: NCT03386110
Title: Couples Health Project: Couples-based Intervention to Reduce Drug Use and HIV Transmission Risk
Acronym: CHP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hunter College of City University of New York (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Tyrel Starks, Associate Professor of Psychology, Hunter College of City University of New York
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R34DA043422 (NIH); R34DA043422 (NIH)
Record Dates: First submitted 2017-12-21; First posted 2017-12-29 (Actual); Results first posted 2021-08-19 (Actual); Last update posted 2021-08-19 (Actual); Status verified 2021-07

CONDITIONS: Risk Behavior; Drug Use; Sex, Anal
Keywords: Couples; MSM; HIV; Drug Use
MeSH Terms: conditions — Risk-Taking; Sexual Behavior | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Couples Health Project (CHP) (Experimental): The CHP intervention is a three session intervention that occurs once a week for three weeks. The CHP intervention will be delivered by MI-trained mental health counselors. The CHP intervention is comprised of 3 sessions. 25 couples will be allocated to this arm.
  Interventions: Behavioral: Couples Health Project (CHP)
- Education (Active Comparator): The Education intervention is a attention-matched control three-session intervention that occurs once a week for three weeks. The education intervention will be delivered by trained health educators. The education intervention is comprised of 3 sessions. 25 couples will be allocated to this arm.
  Interventions: Behavioral: Education

INTERVENTIONS:
Behavioral: Couples Health Project (CHP) — The CHP intervention focuses on addresses drug use and HIV transmission risk by enhancing dyadic communication skills and motivation to work towards shared health goals. The last session of the CHP intervention consists of a Couples HIV Testing and Counseling (CHTC) session.
  Arms: Couples Health Project (CHP)
Behavioral: Education — The Education intervention consists of a 3-session health education intervention that addresses sexual risk and substance use through a lecture and question and answer format with a male couple. Additionally, the last session of the education intervention consists of a Couples HIV Testing and Counseling (CHTC) session.
  Arms: Education

SUMMARY:
This project tests the feasibility, acceptability, and preliminary efficacy of the Couples Health Project (CHP). CHP is a brief (3-session) couples-based Motivational Interviewing intervention which addresses drug use and sexual HIV transmission risk among partnered HIV negative YMSM (ages 18-29). The proposed project includes a randomized controlled trial (RCT) involving 50 couples who are randomized to complete either the CHP intervention or an attention-matched education control condition.

DETAILED DESCRIPTION:
This study aims to evaluate a couples-based intervention with an integrated focus on drug use and HIV prevention, including uptake of and adherence to PrEP. The investigators will recruit a sample of 50 couples (n = 100 individuals)

Recruitment occurs using a mix of in-person and Internet recruitment. Outreach workers will visit bars and events in the New York City area to recruit participants. Also, information on our project will be posted on social media sites (e.g.,Facebook, Grindr, Scruff). Interested individuals will complete a brief online screener to assess eligibility.

A telephone screener will be conducted with participants who are preliminarily eligible based upon online screener responses. Participants who are eligible based upon telephone screening responses will be sent two emails. The first contains a link for them to access the baseline online survey. The second email is for them to forward to their partner. It provides information which introduces the study to the recruited partner and a link to the baseline survey online. If participants indicate intimate partner violence (IPV) on the online baseline survey, participants will be rendered ineligible. Only the participant that indicated experiencing IPV will be given a list of local referrals to access IPV-related services.

An in-person baseline assessment appointment will be scheduled after both participants have completed the online survey. If participants come to the research site alone, they will need to reschedule the appointment when both partners can attend.

The in-person baseline assessment appointment consists of four components; written consenting, a computer-assisted self interview (CASI), a timeline follow back interview, and biological testing.

Written consent is obtained with each participant individually in separate rooms. Participants additionally complete a computer-assisted self interview (CASI) independently. After this, participants will independently complete a TFLB.

TLFB is a semi-structured interview to collect retrospective event-level data on drug use, sexual behavior and PrEP adherence (for those on PrEP) in the past 30 days. Participants complete the survey and TLFB independently in a different room, without their partner.

The final part of the in-person baseline assessment consists of biological testing for STI (gonorrhea & chlamydia via urinalysis and rectal swabs), drug testing via 5-panel fingernail drug assay via finger or toe nail clippings. Drugs tested are 5 major drugs: Amphetamines, Cannabinoids, Cocaine, Opiates, and Phencyclidine (PCP).

After the baseline assessment, participants will be randomized to receive their first CHP or Education session, of which the first session will occur immediately following their baseline assessment. The study will employ a stratified randomization procedure using an algorithm via Qualtrics. Couples will be randomized using three couple-level criteria. Couples will be randomized based on relationship length difference (less than 2 years versus 2 or more), age difference (less than 3 years versus 3 or more), and racial difference (both white versus all others combinations). Each of the intervention arms consists of 3 sessions that occur once a week for three consecutive weeks.

For Session 3 of the experimental and control conditions, participants complete a Couples HIV Testing and Counseling (CHTC) session that involves a rapid HIV testing for couples. HIV testing is done via the Alere Determine HIV-1/2 Ag/Ab Combo blood test. The couple undergo HIV testing together and receive the results together.

All participants complete a 1-month, 3-month, and 6-month follow ups. Follow-up appointments are scheduled with each participant independently (not as a couple). For the 1 month follow up (post baseline assessment), participants will complete an online survey at home for which participants are instructed to take this survey independent from their partner. At the 3 month follow up (post baseline assessment), participants complete a survey with a TLFB and Fingernail specimen collection for drug use at the research office. At the 6 month follow up (post baseline assessment), participants complete a survey with a TLFB and biological specimen collection to test drug use via fingernail sample and Gonorrhea & Chlamydia for STI testing (Urinalysis and Rectal swabs) at the research offices.

ELIGIBILITY:
Inclusion Criteria:

* At least one member of the couple must be 18 to 29 years of age
* Both members assigned male gender at birth and currently identify as male
* At least one member of the couple reports an HIV-negative serostatus
* Couple has been together for at least 3 months
* The use of at least one of the following substances in the past 30 days (only one partner): marijuana, cocaine/crack, amphetamines, ecstasy, GHB, ketamine, nitrates, prescriptionn drug misuse
* At least one member of the couple, in the past 30 days, had condomless anal sex (CAS) with a casual partner and/or CAS with a non-monogamous or serodiscordant main partner.
* Both members must be able to communicate in English
* Both members must reside in the NYC metro area

Exclusion Criteria:

* Either member of the couple reports IPV, which is defined as serious physical or sexual violence that occurs outside the context of consensual bondage or sado-masochistic sexual play, which results in concerns of safety.
* Inconsistencies between information provided in the eligibility screener and the in-person meeting or any issues that might hinder participation. The couple may also be deemed ineligible if participant responses are sufficiently inconsistent to call into question the validity of their individual responses
* The couple reports a sero-concordant HIV-positive serostatus
* Unstable, serious psychiatric symptoms (assessed at Baseline)
* Currently suicidal/homicidal
* Evidence of gross cognitive impairment

Ages: 18 Years to 29 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Eligibility is based on self-identification of a male birth gender and current self-identification of a male gender identity of both parts of the couple.
Enrollment: 100 (Actual)
Dates: Start 2018-03-06 (Actual); Primary Completion 2020-09-14 (Actual); Study Completion 2020-09-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tyrel J Starks, PhD, Principal Investigator — Hunter College of City University of New York
Locations (1):
- Center for HIV Educational Studies and Training, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
A databank may be used to share data consistent with the NIH resource sharing agreement. The requester will contact the PI of the study and the PI will contact the CUNY Office for Research Compliance per university guidelines for data sharing.

REFERENCES:
- [Background] Parsons JT, Lelutiu-Weinberger C, Botsko M, Golub SA. A randomized controlled trial utilizing motivational interviewing to reduce HIV risk and drug use in young gay and bisexual men. J Consult Clin Psychol. 2014 Feb;82(1):9-18. doi: 10.1037/a0035311. Epub 2013 Dec 23. PMID 24364800
- [Derived] Starks TJ, Adebayo T, Kyre KD, Millar BM, Stratton MJ Jr, Gandhi M, Ingersoll KS. Pilot Randomized Controlled Trial of Motivational Interviewing with Sexual Minority Male Couples to Reduce Drug Use and Sexual Risk: The Couples Health Project. AIDS Behav. 2022 Feb;26(2):310-327. doi: 10.1007/s10461-021-03384-9. Epub 2021 Jul 23. PMID 34297275
- [Derived] Starks TJ, Feldstein Ewing SW, Lovejoy T, Gurung S, Cain D, Fan CA, Naar S, Parsons JT. Adolescent Male Couples-Based HIV Testing Intervention (We Test): Protocol for a Type 1, Hybrid Implementation-Effectiveness Trial. JMIR Res Protoc. 2019 Jun 7;8(6):e11186. doi: 10.2196/11186. PMID 31199341

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We used an index participant approach to recruit couples. Online recruitment included advertisements on websites and geosocial networking apps for gay, bisexual, trans, and queer people seeking out sexual partners. Also, staff attended bars, nightclubs, and other social events for these populations in the NYC metro area to screen. Through June 2019, eligible index participants were contacted by phone to complete a study specific screener. This was converted to an online survey in July 2019.
Groups:
- Couples Health Project (CHP): Participants who received the intervention condition, CHP
- Education: Participants who received the attention-matched Education control
Period: Overall Study
Arm/Group | Couples Health Project (CHP) | Education
Started | 56 | 44
Completed | 41 | 38
Not Completed | 15 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Couples Health Project (CHP) | Education | Total
Number analyzed (Participants) | 56 | 44 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 56 | 44 | 100
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.7 (6.17) | 28.05 (6.10) | 28.41 (6.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 56 | 44 | 100
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race & Ethnicity: White/European | 33 | 25 | 58
  Race & Ethnicity: Black/African American | 5 | 6 | 11
  Race & Ethnicity: Latino | 11 | 11 | 22
  Race & Ethnicity: Other | 7 | 2 | 9
Region of Enrollment [Number; unit: participants]
  United States | 56 | 44 | 100
HIV Status [Count of Participants; unit: Participants] — HIV status of each member of the couple was assessed (self-report for those reporting an HIV-positive status, and verified by HIV test for those reporting an HIV-negative status)
  Participants
    HIV-negative | 51 | 39 | 90
    HIV-positive | 5 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: Illicit Drug Use
Description: The self-reported number of illicit drug use instances (not including marijuana) in the past 30 days
Time Frame: Baseline, 3-month follow-up; 6-month follow-up
Population: Intent-to-treat population (assigned to either the CHP intervention or Education Control)
Measure: Mean (Standard Deviation); unit: Days (in the past 30 days)
Arm/Group | Couples Health Project (CHP) | Education
Number analyzed (Participants) | 56 | 44
Days (in the past 30 days)
  Use at Baseline | 3.36 (8.46) | 0.84 (2.34)
  Use at 3-month follow-up | 3.13 (8.41) | 0.73 (1.37)
  Use at 6-month follow-up | 1.17 (3.79) | 0.58 (1.24)
Statistical Analysis 1: Comparison: Couples Health Project (CHP) vs Education; Multi-level models tested whether treatment condition predicted outcome at 3-month follow-up, and controlled for the nesting of participants within couples; Test type: Superiority; p = 0.08, Mixed Models Analysis; Model testing whether condition predicted illicit drug use at 3-months; Risk Ratio, log = 1.19, 95% CI 2-sided [-0.15 to 2.54]
Statistical Analysis 2: Comparison: Couples Health Project (CHP) vs Education; Multi-level models tested whether treatment condition predicted outcome at 6-months, and controlled for the nesting of participants within couples; Test type: Superiority; p = 0.25, Mixed Models Analysis; Model testing whether condition predicted illicit drug use at 6-months; Risk Ratio, log = 0.70, 95% CI 2-sided [-0.49 to 1.89]
Statistical Analysis 3: Comparison: Couples Health Project (CHP) vs Education; Moderation analysis in 3-month follow-up data. The hypothesis that baseline frequency may moderate the effects of treatment at 3-months was evaluated using models incorporating participants' baseline report of the outcome (actor) as well as their partners' report (partner) at Level 1. Interactions among actor and partner baseline scores and treatment condition were also included at Level 1. Additionally, the model controlled for the nesting of participants within couples; Test type: Superiority; p = 0.007, Mixed Models Analysis; Three-way interaction model testing whether baseline use (actor and partner) moderated the effect of condition on illicit drug use at 3-months; Risk Ratio, log = 1.79, 95% CI 2-sided [0.49 to 3.09]
Statistical Analysis 4: Comparison: Couples Health Project (CHP) vs Education; Moderation analysis in 6-month follow-up data. The hypothesis that baseline frequency may moderate the effects of treatment at 6-months was evaluated using models incorporating participants' baseline report of the outcome (actor) as well as their partners' report (partner) at Level 1. Interactions among actor and partner baseline scores and treatment condition were also included at Level 1. Additionally, the model controlled for the nesting of participants within couples; Test type: Superiority; p = 0.71, Mixed Models Analysis; Three-way interaction model testing whether baseline use (actor and partner) moderated the effect of condition on illicit drug use at 6-months; Risk Ratio, log = -0.36, 95% CI 2-sided [-2.26 to 1.53]

2. Primary Outcome: Number of HIV Transmission Risk Events
Description: The self-reported number of events of condomless anal sex (CAS) with casual partners in the past 30 days
Time Frame: 6 months
Population: Intent-to-treat population (assigned to either the CHP intervention or Education Control)
Measure: Mean (Standard Deviation); unit: Events in the past 30 days
Arm/Group | Couples Health Project (CHP) | Education
Number analyzed (Participants) | 56 | 44
Events in the past 30 days
  Events at Baseline | 1.68 (2.78) | 1.68 (2.34)
  Events at 3-month follow-up | 2.13 (3.61) | 1.49 (3.70)
  Events at 6-month follow-up | 0.88 (1.66) | 1.05 (1.82)
Statistical Analysis 1: Comparison: Couples Health Project (CHP) vs Education; Multi-level models tested whether treatment condition predicted outcome at 3-months, and controlled for the nesting of participants within couples; Test type: Superiority; p = 0.36, Mixed Models Analysis; Model testing whether condition predicted CAS events at 3-months; Risk Ratio, log = 0.36, 95% CI 2-sided [-0.65 to 1.37]
Statistical Analysis 2: Comparison: Couples Health Project (CHP) vs Education; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.63, Mixed Models Analysis; Model testing whether condition predicted CAS events at 6-months; Risk Ratio, log = -0.18, 95% CI 2-sided [-1.15 to 0.78]
Statistical Analysis 3: Comparison: Couples Health Project (CHP) vs Education; [analysis description as in outcome 1, analysis 3]; Test type: Superiority; p = 0.42, Mixed Models Analysis; Three-way interaction model testing whether baseline rates of CAS (actor and partner) moderated the effect of condition on CAS events at 3-months; Risk Ratio, log = -0.54, 95% CI 2-sided [-1.85 to 0.77]
Statistical Analysis 4: Comparison: Couples Health Project (CHP) vs Education; [analysis description as in outcome 1, analysis 4]; Test type: Superiority; p = 0.02, Mixed Models Analysis; Three-way interaction model testing whether baseline rates of CAS (actor and partner) moderated the effect of condition on CAS events at 6-months; Risk Ratio, log = -1.70, 95% CI 2-sided [-3.14 to -0.27]

3. Secondary Outcome: Marijuana Use
Description: The self-reported number of marijuana drug use instances in the past 30 days
Time Frame: 6 months
Population: Intent-to-treat population (assigned to either the CHP intervention or Education Control)
Measure: Mean (Standard Deviation); unit: days out of 30
Arm/Group | Couples Health Project (CHP) | Education
Number analyzed (Participants) | 56 | 44
days out of 30
  Use at Baseline | 9.61 (11.93) | 7.02 (10.24)
  Use at 3-month follow-up | 9.62 (11.83) | 5.95 (10.24)
  Use at 6-month follow-up | 10.00 (12.43) | 7.89 (11.75)
Statistical Analysis 1: Comparison: Couples Health Project (CHP) vs Education; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.15, Mixed Models Analysis; Model testing whether condition predicted marijuana use at 3-months; Risk Ratio, log = 0.48, 95% CI 2-sided [-0.18 to 1.44]
Statistical Analysis 2: Comparison: Couples Health Project (CHP) vs Education; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.50, Mixed Models Analysis; Model testing whether condition predicted marijuana use at 6-months; Risk Ratio, log = 0.24, 95% CI 2-sided [-0.44 to 0.92]
Statistical Analysis 3: Comparison: Couples Health Project (CHP) vs Education; Moderation analysis in 3-month follow-up data. The hypothesis that baseline frequency may moderate the effects of treatment was evaluated using models incorporating participants' baseline report of the outcome (actor) as well as their partners' report (partner) at Level 1. Interactions among actor and partner baseline scores and treatment condition were also included at Level 1. Additionally, the model controlled for the nesting of participants within couples; Test type: Superiority; p = 0.910, Mixed Models Analysis; Three-way interaction model testing whether baseline use moderated the effect of condition on marijuana use at 3-months; Risk Ratio, log = -0.02, 95% CI 2-sided [-0.34 to 0.31]
Statistical Analysis 4: Comparison: Couples Health Project (CHP) vs Education; Moderation analysis in 6-month follow-up data. The hypothesis that baseline frequency may moderate the effects of treatment was evaluated using models incorporating participants' baseline report of the outcome (actor) as well as their partners' report (partner) at Level 1. Interactions among actor and partner baseline scores and treatment condition were also included at Level 1. Additionally, the model controlled for the nesting of participants within couples; Test type: Superiority; p = 0.11, Mixed Models Analysis; Risk Ratio, log = 0.34, 95% CI 2-sided [-0.07 to 0.75]

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Couples Health Project (CHP) | Education
All-Cause Mortality (participants affected / at risk) | 0/56 | 0/44
Serious Adverse Events (participants affected / at risk) | 0/56 | 0/44
Other Adverse Events (participants affected / at risk) | 0/56 | 0/44

LIMITATIONS AND CAVEATS:
This was a pilot study with modest sample size intended to test preliminary efficacy and provide effect size estimates necessary to plan a larger trial. Results warrant replication in research with larger sample size. The sample was recruited from a large urban center and may not be representative of the wider U.S. population of partnered sexual minority men. Due to COVID, the collection of follow-up STI specimen data was curtailed, diminishing our ability to test associations with this outcome.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-05-15): https://cdn.clinicaltrials.gov/large-docs/10/NCT03386110/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-01): https://cdn.clinicaltrials.gov/large-docs/10/NCT03386110/SAP_001.pdf